CLINICAL TRIAL: NCT01133951
Title: Helicobacter Pylori Eradication to Prevent Gastric Cancer in a High-Risk Population of China: A Randomized Controlled Trial
Brief Title: Helicobacter Pylori Eradication to Prevent Gastric Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jie-Jun Wang (Other)
Responsible Party: Sponsor-Investigator, Jie-Jun Wang, MD, Second Military Medical University
Organization: Second Military Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SMMU20100501
Record Dates: First submitted 2010-05-28; First posted 2010-05-31 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Helicobacter Infections; Stomach Neoplasms
Keywords: Helicobacter Infections; Helicobacter pylori; Drug Therapy; Precancerous Conditions; Stomach Neoplasms; Incidence
MeSH Terms: conditions — Helicobacter Infections; Stomach Neoplasms; Precancerous Conditions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OAC triple therapy (Experimental)
  Interventions: Drug: OAC triple therapy
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OAC triple therapy — Omeprazole, 20mg, amoxicillin, 1000mg, and clarithromycin, 500mg, all twice a day for 2 weeks.
  Arms: OAC triple therapy
Drug: Placebo — Omeprazole placebo, amoxicillin placebo, and clarithromycin placebo, all twice a day for 2 weeks.
  Arms: Placebo

SUMMARY:
Gastric cancer is the fourth most common type of cancer and the second leading cause of cancer-related death in the world. In China, more than 390,000 new patients are diagnosed with gastric cancer and more than 300,000 patients are killed by the terrible disease annually. Although gastric cancer has a multifactorial etiology, infection with H. pylori is highly associated with gastric carcinogenesis. Therefore, eradication of H. pylori infection appears to reduce the risk of gastric cancer. However, several recent controlled interventional trials by H. pylori eradication to prevent gastric cancer have yielded disappointing results. The exact effect of H.pylori eradication on prevention of gastric cancer is unclear up to now. To clarify this problem, the investigators conducted a prospective, randomized, double-blind, placebo-controlled, population-based study to determine whether H pylori eradication would reduce the incidence of gastric cancer in a high-risk population in China.

ELIGIBILITY:
Inclusion Criteria:

* Healthy registered inhabitants from 10 villages in a high-risk county of gastric cancer in China
* Age 30-59 years
* A willingness to participate in the study as indicated by written informed consent

Exclusion Criteria:

* Severe concomitant illness (eg, severe hypertension, coronary heart disease, diabetes mellitus, stroke, asthma, liver cirrhosis, tuberculosis, infectious hepatitis, and cardiac, respiratory, hepatic, or renal insufficiency)
* Patients with epilepsy or severe mental illness
* Previous diagnosis of cancer
* A history of esophageal or gastric surgery
* Drug abuse and drug dependence
* Allergic to omeprazole, amoxicillin, or clarithromycin
* Pregnant and lactating women
* Previous history of H pylori eradication treatment
* A negative 13C-urea breath test (UBT)
* A definite indication of H. pylori eradication (eg, gastric or duodenum ulcer)
* Dysplasia or carcinoma lesions are found in esophageal or gastric histopathological examination
* Other factors or conditions might influence the results of study

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3000 (Actual)
Dates: Start 2010-06; Primary Completion 2012-01 (Actual); Study Completion 2032-05 (Estimated)

PRIMARY OUTCOMES:
Gastric cancer incidence | 10 years
  The incidence of gastric cancer in the two groups

SECONDARY OUTCOMES:
Histopathological changes | 10 years
  The histopathological changes of atrophic gastritis or intestinal metaplasia in the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Jie J Wang, M.D., Study Chair — Shanghai Changzheng Hospital affiliated to Second Military Medical University; Xi Wang, M.D., Principal Investigator — Shanghai Changzheng Hospital affiliated to Second Military Medical University
Locations (1):
- Zhao-Lai Hua M.D., Yangzhong, Jiangsu, China